CLINICAL TRIAL: NCT02046811
Title: Reducing Skin Cancer Risk in Childhood Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Cancer Institute (NCI) (NIH); St. Jude Children's Research Hospital (Other); Dana-Farber Cancer Institute (Other); Memorial Sloan Kettering Cancer Center (Other); Emory University (Other)
Responsible Party: Principal Investigator, Alan Geller, RN, MPH, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1R01CA175231 (NIH); R01CA175231 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Skin Neoplasms
Keywords: Skin neoplasms; Radiation; Screening; Self-examination; Comparative effectiveness research; Dermoscopy
MeSH Terms: conditions — Skin Neoplasms; Self-Examination | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patient activation and education (Experimental): Patient activation and education (PAE)
  Interventions: Behavioral: Patient activation and education (PAE)
- PAE plus physician activation (Experimental): PAE plus physician activation (PAE + MD)
  Interventions: Behavioral: PAE plus physician activation (PAE + MD)
- PAE, MD, plus teledermoscopy (Experimental): PAE physician activation, plus teledermoscopy (PAE +MD +TD)
  Interventions: Behavioral: PAE physician activation, plus teledermoscopy (PAE +MD +TD)

INTERVENTIONS:
Behavioral: Patient activation and education (PAE) — Text messaging and web-based tutorials for a 12-month duration (a website and smartphone interface)
  Arms: Patient activation and education
Behavioral: PAE plus physician activation (PAE + MD) — Text messaging and web-based tutorials for a 12-month duration (a website and smartphone interface), physician activation/educational materials about: (1) survivors' increased skin cancer risk; (2) the benefits of and the skills needed to conduct full-body skin exams; and (3) the importance of recommending routine SSE to patients
  Arms: PAE plus physician activation
Behavioral: PAE physician activation, plus teledermoscopy (PAE +MD +TD) — Text messaging and web-based tutorials for a 12-month duration (a website and smartphone interface), physician activation/educational materials about: (1) survivors' increased skin cancer risk; (2) the benefits of and the skills needed to conduct full-body skin exams; and (3) the importance of recommending routine SSE to patients, and participant receipt of a dermoscopic lens
  Arms: PAE, MD, plus teledermoscopy

SUMMARY:
The objective of this study is to determine the impact of a 12-month patient activation and education intervention on skin cancer early detection practices among childhood cancer survivors treated with radiation. This randomized controlled trial uses a three-group design.

Our specific aims are to: (1) Determine the impact of a Patient Activation and Education intervention with and without physician activation and teledermatology on skin cancer early detection practices, (2) Determine the impact of the intervention on time to diagnosis, and (3) Estimate the cost and cost-effectiveness of the intervention as a secondary outcome.

DETAILED DESCRIPTION:
There are currently more than 420,000 Americans who are long-term survivors of childhood and adolescent cancer. While these groups have greatly benefited from recent medical advances, primarily increasing overall survival rates, treatment advances have come at a cost. It is now clear that childhood radiation therapy has caused survivors to be at extremely high risk for non-melanoma skin cancer (NMSC) and increased risk of melanoma. Early detection is crucial to reduce the morbidity caused by NMSCs and the morbidity and mortality incurred due to melanoma. Both patient and provider action are needed to detect and treat early skin cancers and to find new solutions to ensure expedited follow-up care and treatment, especially among those who live where they have little access to dermatologists.

The objective of this study is to determine the impact of a 12-month patient activation and education intervention on skin cancer early detection practices among childhood cancer survivors treated with radiation. All participants will receive text messages encouraging them to examine their skin and request physician examinations while concurrently driving them to a study website that provides education related to the associated skills, and reinforces and expands the text messages. To reduce skin cancers among this young and dispersed patient population, this study will address several key issues: (1) how to provide patients with the skills needed to conduct effective skin self-examinations; 2) how to prompt action from patient's physicians when worrisome moles and lesions are found; and 3) how to ensure rapid access to dermatologic exams, which in some parts of the US can take weeks or months to schedule.

ELIGIBILITY:
Inclusion Criteria:

* treated with radiation for a childhood cancer
* have a regular healthcare provider whom he/she has seen in the previous 2 years, or plans to see in the next year
* have a phone that can receive text messages
* have access to a dermlite compatible smartphone or tablet

Exclusion Criteria:

* personal history of a skin cancer diagnosis

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Patient thorough skin self-examination (TSSE) | 18 months
  Self-report of patient thorough skin self-examination (TSSE) will be defined as performing at least one TSSE during the 2 months prior to the 18-month follow-up assessment.

SECONDARY OUTCOMES:
Completion of a physician skin exam | 18 months
  Completion of a physician skin exam will be assessed by participant report and chart review.
Shorter time interval to diagnostic visit | 18 months
  A shorter time interval between the first finding of a suspect lesion after randomization and a diagnostic visit will be assessed by participant report and chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Geller, RN, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geller AC, Coroiu A, Keske RR, Haneuse S, Davine JA, Emmons KM, Daniel CL, Gibson TM, McDonald AJ, Robison LL, Mertens AC, Elkin EB, Marghoob A, Armstrong GT. Advancing Survivors Knowledge (ASK Study) of Skin Cancer Surveillance After Childhood Cancer: A Randomized Controlled Trial in the Childhood Cancer Survivor Study. J Clin Oncol. 2023 Apr 20;41(12):2269-2280. doi: 10.1200/JCO.22.00408. Epub 2023 Jan 9. PMID 36623247
- [Derived] Daniel CL, Armstrong GT, Keske RR, Davine JA, McDonald AJ, Sprunck-Harrild KM, Coleman C, Haneuse SJ, Mertens AC, Emmons KM, Marghoob AA, Elkin EB, Dusza SW, Robison LL, Geller AC. Advancing Survivors' Knowledge (ASK) about skin cancer study: study protocol for a randomized controlled trial. Trials. 2015 Mar 24;16:109. doi: 10.1186/s13063-015-0637-x. PMID 25873142